CLINICAL TRIAL: NCT04634955
Title: Comparison of Intravascular Incidence With Different Fluoroscopic Approach Method During S1 Trasnforaminal Injection
Brief Title: S1 Transforaminal Injection and Vascular Incidence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Principal Investigator, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-08-028
Record Dates: First submitted 2020-11-10; First posted 2020-11-18 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Inadvertent Arterial Puncture
Keywords: intravascular injection transforaminal injection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S1 transforaminal injection with oboique view (Active Comparator): S1 transforaminal injection with oblique fluoroscopic view
  Interventions: Procedure: tranforaminal epidural injection
- S1 transforaminal injection with AP view (Active Comparator): S1 transforaminal injection with anteroposterior fluoroscopic view
  Interventions: Procedure: tranforaminal epidural injection

INTERVENTIONS:
Procedure: tranforaminal epidural injection — tranforaminal epidural injection which is performed by fluoroscopic guidance

SUMMARY:
Intravascular incidence during S1 transforaminal injection is known to be higher than lumbar injection. Its incidence is reported to be 15~25%.

This study was aimed to see if there is any benefit of reducing the intravasuclar injection rate when S1 transforaminal injection was performed by different fluorosopic approach.

DETAILED DESCRIPTION:
Fluorosocpically guided transforaminal epidural steroid injection is a popular interventional procedure that is effective in radicular pain conditions such as herniated interverebral disc, spinal stenosis and failed back surgery syndrome.

The incidence of inadvertent intravascular needle injection during lumbar transforaminal injection is reported as from 9.9% to 30.8%. In particular, S1 intravascular injection rate is more frequent than at the lumbar level.

Previous study reported that guiding the needle toward the S1 foramen using the S1 scotty dog image as a bony landmark, not in the classic way, but in an oblique fluoroscopic view, during L5 and S1 transforaminal epidural steroid injection, can save procedure time and reduce the risk of radiation exposure.

In this stidy, the investigators aimed to compare the incidence of intravascular injection rate by anteroposterior and oblique view approaches for S1 transforaminal epidural steroid injection. In addition, the investigators also compared the procedure time and radiation exposure between two approach method.

ELIGIBILITY:
Inclusion Criteria:

* spinal stenosis
* herniated intervertebral disc
* failed back surgery syndrome

Exclusion Criteria:

* coagulopathy
* infection

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
intravascular incidence | 15 minutes after the completion of the intervention
  intravascular injection rate

SECONDARY OUTCOMES:
procedure time | 15 minutes after the completion of the intervention
  procedure time
radiation dose | 15 minutes after the completion of the intervention
  radiation dose

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hee Hong, PhD, Principal Investigator — Keimyung University
Locations (1):
- Hong ji HEE, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No